CLINICAL TRIAL: NCT03673020
Title: Phase 1a First-in-Human Study of Safety and Tolerability of ASV® AGEN2017 With QS-21 Stimulon® Adjuvant as a Single Agent in Subjects With Solid Tumor at Risk of Relapse Undergoing Observation as SOC Following Complete Surgical Resection
Brief Title: Phase 1a Study to Evaluate Immunogenicity of ASV®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-610-01
Record Dates: First submitted 2018-09-11; First posted 2018-09-17 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumor, Adult
Keywords: Vaccine; Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ASV® AGEN2017 (Experimental): ASV® AGEN2017 + QS-21 Stimulon® Adjuvant Vaccine
  Interventions: Biological: ASV® AGEN2017 + QS-21 Stimulon® adjuvant

INTERVENTIONS:
Biological: ASV® AGEN2017 + QS-21 Stimulon® adjuvant — Neoantigen Vaccine

SUMMARY:
This is an open-label Phase 1a First-in-Human Study to determine Safety and Tolerability of ASV® AGEN2017 with QS-21 Stimulon® Adjuvant as a Single Agent in Subjects With Tumors at Risk of Relapse Undergoing Observation as Standard of Care Following Complete Surgical Resection.

DETAILED DESCRIPTION:
This is a Phase 1a study to evaluate neoantigen vaccine, AutoSynVax (ASV®) AGEN2017 in subjects with resected solid tumors, no evidence of disease (NED), and with an estimated life expectancy of ≥12 months from the time tissue has been submitted for vaccine manufacture. A minimum of 3 subjects will be enrolled to receive every two weeks subcutaneous injection of AGEN2017 + QS-21 adjuvant.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, written informed consent.
2. Age ≥18 years.
3. Diagnosis of solid cancer that has been completely resected, NED, and eligible for observation only as SOC yet remain at risk of relapse per Investigator discretion. These include subjects diagnosed with malignant melanoma, non-small cell lung cancer, bladder cancer, colorectal cancer, breast cancer, renal cancer, head and neck cancer, cervical cancer, and soft tissue sarcoma.
4. Life expectancy ≥12 months from the time of consent.
5. Available fresh tissue from surgical excision. If fresh tissue is not available, formalin-fixed paraffin-embedded archival tissue may be used. The modality of the biopsy (e.g., endobronchial ultrasound, bronchoscopic, computed-tomography-guided needle biopsy) is not specified; however, core biopsy and fine needle aspiration are acceptable as long as the biopsy can be prepared as a cell block in paraffin-embedded tissue.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Adequate bone marrow function, as measured from studies of peripheral blood (absolute neutrophil count ≥1,500/mm3, absolute lymphocyte count ≥500/mm3, platelet count 50,000/mm3, hemoglobin >8.0 mg/dL).
8. Adequate cardiac function (New York Heart Association class ≤II).
9. Female subjects of childbearing potential must have a negative serum pregnancy test at the screening and pretreatment visits, and prior to first dose of study medication. Non-childbearing potential (other than by medical reasons) is defined as 1 of the following:

   1. ≥45 years of age and amenorrheic for >1 year by self-report.
   2. Amenorrheic for >2 years without a hysterectomy and oophorectomy, and follicle-stimulating hormone value in the postmenopausal range upon screening evaluation.
   3. Status post-hysterectomy, -oophorectomy, or -tubal ligation. If of childbearing potential, female subjects must be willing to use adequate birth control during the study, starting with the screening visit through 120 days after the last dose of study therapy.

   Male subjects with a female partner(s) of childbearing potential must agree to use a condom throughout the trial, starting with the screening visit through 120 days after the last dose of study therapy. Male subjects with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

   Note: Abstinence is acceptable for both female and male subjects if this is the subject's established and preferred contraception method.
10. Subject is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Subjects must not have received anticancer medications or investigational drugs within the following intervals before first dose of study drug:

   1. ≤14 days for chemotherapy, targeted small molecule therapy, anticancer hormone therapy, or radiation therapy, with the following exceptions:

      * Bisphosphonates and denosumab are permitted.
      * Novel imaging agents that have Phase 1 safety data and have not demonstrated therapeutic activity are permitted.
      * Physiologic steroid replacement for adrenal insufficiency (e.g., <10 mg prednisone per day) is permitted.
      * Prophylactic use of inhaled or topical corticosteroid or short course of intravenous systemic corticosteroid (≤3 days) for radiographic procedures is permitted.
      * Use of physiologic corticosteroid replacement therapy must be approved by the medical monitor.
   2. ≤28 days for prior cancer immunotherapy.
   3. ≤28 days for prior monoclonal antibody used for anticancer therapy, with the exception of denosumab.
   4. ≤7 days for immunosuppressive treatment for any reason. Systemic corticosteroids are not allowed except as defined above.
   5. e. ≤28 days before first dose of study drug for all other investigational study drugs or devices.

   Note: Washout is applicable to the screening visit only, and not applicable prior to the first dose of study drug. Subjects are not to receive anti-cancer therapies from date of consent through the post treatment visit (end of treatment or final safety visit).
2. Diagnosis of clinically significant immunodeficiency (as defined by the principal investigator), or actively receiving or potentially needing any form of immunosuppressive therapy within 7 days prior to the first dose of study drug until the end of the trial.
3. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator or medical monitor.
4. Uncontrolled intercurrent illness, including but not limited to uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or social situations that would limit compliance with study requirements in the opinion of the treating investigator or medical monitor.
5. History of intolerance or allergic reactions attributed to compounds of similar chemical or biologic composition to AGEN2017 or QS-21 adjuvant.
6. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergence Adverse Events (Safety and Tolerability) | 1 Year
  Assessed by monitoring the frequency, duration, and severity of drug-related AEs by completing physical examinations and clinical evaluations; evaluating changes in vital signs; and laboratory blood and urine sample evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.
Locations (1):
- School of Medicine at the University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No